CLINICAL TRIAL: NCT04989660
Title: Phenol Neurolysis of Genicular Nerves for Osteoarthritic Knee Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-1154-21
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Knee; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Phenol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): 6% aqueous phenol, 1.5 mL per target site
  Interventions: Drug: 6% aqueous phenol
- Placebo Group (Placebo Comparator): Isotonic saline, 1.5 mL per target site
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: 6% aqueous phenol — 1.5 mL of 6% aqueous phenol will be injected at each target genicular nerve under ultrasound guidance.
  Other Names: Phenol
  Arms: Treatment Group
Drug: Isotonic saline — 1.5 mL of isotonic saline will be injected at each target genicular nerve under ultrasound guidance.
  Arms: Placebo Group

SUMMARY:
As the aging and obese populations continue to increase, there is a rapidly growing number of people at risk for knee osteoarthritis. Treatment typically starts conservatively with analgesics, physical therapy, and bracing. Intra-articular injections with corticosteroids and/or viscosupplementation may also be utilized in those with persistent knee pain. Genicular nerve radiofrequency ablation (GNRFA) is an increasingly employed procedure for refractory osteoarthritic knee pain with promising efficacy for pain relief. However, due to its reliance on expensive equipment, additional staff, and need for specialized rooms (eg. fluoroscopy suite), GNRFA is a costly procedure with limited availability. Chemical neurolysis is an alternative method of nerve ablation using alcohol or phenol utilized in the management of pain. Recent literature has demonstrated good efficacy for pain relief and function with chemical ablation of the genicular nerves using both alcohol and phenol.

This study is a double-blind, randomized, placebo-controlled pilot study to assess the efficacy of phenol neurolysis of the genicular nerves for pain and function due to refractory osteoarthritic knee pain. We hypothesize that a significant improvement in both pain and function will be observed with chemical neurolysis of the genicular nerves using 6% phenol compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic knee osteoarthritis (Kellgren-Lawrence grade 2-4)
* Knee pain of moderate intensity or greater (NRS of 4 or greater)
* Knee pain for 3 months or longer
* Persistent knee pain despite conservative treatment including oral/topical analgesics, physiotherapy, intra-articular injection with corticosteroid and/or hyaluronic acid

Exclusion Criteria:

* Prior total or partial knee arthroplasty in the knee(s) to be treated
* Prior radiofrequency ablation treatment in the affected knee
* Other rheumatological or connective tissue disease(s) affecting the knee to be treated
* History of bleeding disorder
* Any psychiatric or neurologic disease (eg. dementia, brain injury, etc.) that may preclude reliable reporting of symptoms and response to treatment
* Pregnancy
* Recent treatment with intraarticular hyaluronic acid, platelet-rich plasma, or corticosteroid injections to the affected knee in the past 3 months
* Skin or joint infection in the knee(s) to be treated
* Concomitant radicular pain

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in NRS pain score from baseline | Baseline, 1 month, 3 months, 6 months
  Participants' pain will be measured using the numeric rating scale (0-10) prior to the intervention and at 1 month, 3 months, and 6 months after the intervention. Numeric rating scale ranges from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Change in WOMAC score from baseline | Baseline, 1 month, 3 months, 6 months
  Participants' function as measured by WOMAC will be measured prior to the intervention and at 1 month, 3 months, and 6 months after the intervention. WOMAC score ranges from 0 (best) to 100 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Paul So, MD, Principal Investigator — Kessler Institute for Rehabilitation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No